CLINICAL TRIAL: NCT00311129
Title: A Multicenter Study to Assess the Antitumor Effect and Safety of Fludarabine Phosphate Tablet (SH T 586) in Combination With Rituximab Administered in 6 Treatment Cycles (1 Treatment Cycle: Rituximab 375 mg/m2 iv on Day 1 Along With 5-Consecutive Day Oral Dosing of SH T 586 40 mg/m2/Day From Day 1 to Day 5, Followed by an Observation Period of 23 Days) in Patients With Indolent Lymphoma
Brief Title: Efficacy and Safety Study of SH T 586 in Combination With Rituximab to Treat Low-Grade NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 309123; 91456
Record Dates: First submitted 2006-03-31; First posted 2006-04-05 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma, Low-Grade
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — fludarabine phosphate; Rituximab

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Fludarabine Phosphate (Fludara)
- Arm 2 (Active Comparator)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine Phosphate (Fludara) — Injection of rituximab on Day 1 along with 5-consecutive day oral dosing of fludarabine phosphate from Day 1 to Day 5, followed by an observation period from Day 6 to Day 28 as 1 treatment cycle, 6 cycles will be given. As for patients who has been observed with partial response (PR) or better antitumor effect, any treatment shall not be provided in principle until the status comes to progressive disease (PD)
  Other Names: BAY86-4864
  Arms: Arm 1
Drug: Rituximab — Injection of rituximab on Day 1, followed by an observation period from Day 6 to Day 28 as 1 treatment cycle, 6 cycles will be given. As for patients who has been observed with partial response (PR) or better antitumor effect, any treatment shall not be provided in principle until the status comes to progressive disease (PD)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess the antitumor effect and safety of fludarabine phosphate tablet in combination with rituximab in patient with indolent lymphoma.

DETAILED DESCRIPTION:
As of 29 May 2009, the clinical trial sponsor is Genzyme Corporation. NOTE: This study was originally posted by sponsor Schering AG, Germany, which was subsequently renamed to Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD 20 positive, relapsed/refractory indolent lymphoma. (Regimens of prior chemotherapy are limited to 2; prior rituximab treatments up to 16 times are allowed.)
* Patients with measurable lesions (> 1.5 cm).
* Patients who have not received any treatment for more than 4 weeks after completing previous therapies (6 months in the case of antibody therapies).
* ECOG performance status: 0 - 1
* Patients with adequately maintained organ functions.

Exclusion Criteria:

* Patients with infectious disease, serious complications, serious gastrointestinal symptoms, serious bleeding tendency, serious CNS symptoms, fever </=38 °C, interstitial pneumonia or pulmonary fibrosis, active other malignancies, autoimmune hemolytic anemia or the history of the disease, or glaucoma.
* Patients who are positive for HBs antigen, HCV antibody, or HIV antibody.
* Patients who received G-CSF or transfusion within 1 week before the registration.
* Patients with the history of allergies to purine nucleoside analogue.
* Patients who experienced serious hypersensitivity or anaphylaxis to rituximab or mouse protein-derived products.
* Patients who had ever received prior therapy with fludarabine phosphate injection, pentostatin, cladribine, SH T 586, blood stem cell transplant, or monoclonal antibody therapy other than rituximab to NHL (including radioimmunotherapy).
* Patients who had progressive disease within 6 months of receiving therapy including rituximab.
* Women who are pregnant, of childbearing potential, or lactating.
* Patients who do not agree to practice contraception.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | The best response until the end of 6th treatment cycle

SECONDARY OUTCOMES:
CR rate | CR or CRu until the end of 6th treatment cycles
Progression free survival | Progression or death which comes earlier, observed until 12 weeks after the completion of the treatment in the last patient
Overall survival | Death, observed until 12 weeks after the completion of the treatment in the last patient

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- Japan (7):
  - Nagoya, Aichi-ken
  - Kashiwa-shi, Chiba
  - Isehara-shi, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Hamamatsu, Shizuoka
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Tobinai K, Ishizawa K, Ogura M, Itoh K, Morishima Y, Ando K, Taniwaki M, Watanabe T, Yamamoto J, Uchida T, Nakata M, Terauchi T, Nawano S, Matsusako M, Hayashi M, Hotta T. Phase II study of oral fludarabine in combination with rituximab for relapsed indolent B-cell non-Hodgkin lymphoma. Cancer Sci. 2009 Oct;100(10):1951-6. doi: 10.1111/j.1349-7006.2009.01247.x. Epub 2009 Jun 17. PMID 19594547